CLINICAL TRIAL: NCT02879383
Title: Evaluation of the Effect of Duodenal Mucosal Resurfacing (DMR) Using the Revita System in the Treatment of Type 2 Diabetes (T2D)
Brief Title: Effect of Duodenal Mucosal Resurfacing (DMR) Using the Revita System in the Treatment of Type 2 Diabetes (T2D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-30000
Record Dates: First submitted 2016-08-04; First posted 2016-08-25 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2; Noninsulin-Dependent Diabetes Mellitus
Keywords: Type 2 Diabetes, Revita System, DMR
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMR Procedure (Experimental): Subjects randomized to the DMR procedure are unblinded at 24 weeks and followed for an additional 24 weeks.
  Interventions: Procedure: DMR Procedure
- Sham Procedure (Sham Comparator): Subjects are unblinded at 24 Weeks. Sham subjects to cross over to receive DMR treatment at 24 Weeks and followed up for additional 24 weeks.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Procedure: DMR Procedure — The DMR procedure consists of hydrothermal ablation of the duodenum using the Revita System
  Other Names: DMR; Revita
  Arms: DMR Procedure
Procedure: Sham Procedure — The sham procedure consists of placing the Revita Catheter into the stomach for 30 minutes and then removing it from the patient.
  Arms: Sham Procedure

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of the Fractyl duodenal mucosal resurfacing (DMR) Procedure using the Revita System compared to a sham procedure for the treatment of uncontrolled type 2 diabetes.

Subjects randomized to the DMR procedure are followed per protocol for 48 Weeks. The Sham treatment arm will cross over to receive the DMR treatment at 24 weeks with background medications held constant from 24-48 weeks of follow up.

DETAILED DESCRIPTION:
The study is a multi-center, randomized, prospective, double-blinded (subject and endocrinologist) trial of type 2 diabetes patients sub-optimally controlled on 1 or more oral anti-diabetic medications comparing the Fractyl DMR procedure to sham procedure. Randomization will be 1:1 DMR treatment to sham. All subjects will participate in a 4 week oral anti-diabetic medication run-in period before the index procedure to confirm lack of blood glucose control in conjunction with medication compliance and nutritional counseling. The Sham treatment arm will cross-over to receive the DMR treatment at 24 weeks with background medications held constant 24weeks of follow up after the cross-over DMR procedure. The DMR treatment arm will be managed according to current diabetes standard of care.

Subjects randomized to the DMR procedure are followed per protocol for 48 Weeks. The Sham treatment arm will cross over to receive the DMR treatment at 24 weeks with background medications held constant from 24-48 weeks of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. 28-75 years of age
2. Diagnosed with Type 2 Diabetes and evidence of preserved insulin secretion. Fasting insulin > 7 μU/ mL.
3. Glycated Hemoglobin (HbA1c) of 7.5 - 10.0% (59-86 mmol/mol)
4. Body Mass Index (BMI) ≥ 24 and ≤ 40 kg/m2
5. Currently taking one or more oral glucose lowering medications of which one must be Metformin, with no changes in dose or medication in the previous 12 Weeks prior to study entry
6. Able to comply with study requirements and understand and sign the informed consent

Exclusion Criteria:

1. Diagnosed with Type 1 Diabetes or with a history of ketoacidosis
2. Current use of Insulin
3. Current use of Glucagon-like peptide-1 (GLP-1) analogues
4. Hypoglycemia unawareness or a history of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party-assistance, in the last year)
5. Known autoimmune disease, as evidenced by a positive Anti- Glutamic Acid Decarboxylase (GAD) test, including Celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
6. Active H. pylori infection (Participants with active H. pylori may continue with the screening process if they are treated via medication and re-testing verifies the condition has resolved.)
7. Previous GI surgery that could affect the ability to treat the duodenum such as subjects who have had a Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions
8. History of chronic or acute pancreatitis
9. Known active hepatitis or active liver disease
10. Symptomatic gallstones or kidney stones, acute cholecystitis or history of duodenal inflammatory diseases including Crohn's Disease and Celiac Disease
11. History of coagulopathy, upper gastro-intestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia
12. Use of anticoagulation therapy (such as warfarin) which cannot be discontinued for 7 days before and 14 days after the procedure
13. Use of P2Y12 inhibitors (clopidogrel, pasugrel, ticagrelor) which cannot be discontinued for 14 days before and 14 days after the procedure. Use of aspirin is allowed.
14. Unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during treatment through 4 weeks post procedure phase
15. Taking corticosteroids or drugs known to affect GI motility (e.g. Metoclopramide)
16. Receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
17. Persistent Anemia, defined as Hgb<10 g/dl
18. Estimated Glomerular Filtration Rate (eGFR) or Modified of Diet in Renal Diseae (MDRD) <30 ml/min/1.73m^2
19. Active systemic infection
20. Active malignancy within the last 5 years
21. Not potential candidates for surgery or general anesthesia
22. Active illicit substance abuse or alcoholism
23. Participating in another ongoing clinical trial of an investigational drug or device
24. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD, PhD, Principal Investigator — Gemelli University Hospital, Rome; Jacques Bergman, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (11):
- Belgium (2):
  - Hopital Erasme, Brussels
  - UZ Leuven, Leuven
- Brazil (2):
  - ABC Hospital, São Paulo
  - Hospital das Clinicas da Faculdade de medicina da Universidade de São Paulo, São Paulo
- Italy (2):
  - Policlinico Gemelli (Sacro Cuore), Rome, Lazio
  - Humanitas Research Hospital & Humanitas University Via Manzoni 56, Rozzano, Milan
- Amsterdam University Medical Center, Amsterdam, Netherlands
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow
  - University College London Hospitals, London
  - King's College, Denmark Hill, London
  - Queens Medical Centre campus, Nottingham University Hospitals NHS Trust, Derby Road, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mingrone G, van Baar AC, Deviere J, Hopkins D, Moura E, Cercato C, Rajagopalan H, Lopez-Talavera JC, White K, Bhambhani V, Costamagna G, Haidry R, Grecco E, Galvao Neto M, Aithal G, Repici A, Hayee B, Haji A, Morris AJ, Bisschops R, Chouhan MD, Sakai NS, Bhatt DL, Sanyal AJ, Bergman JJGHM; Investigators of the REVITA-2 Study. Safety and efficacy of hydrothermal duodenal mucosal resurfacing in patients with type 2 diabetes: the randomised, double-blind, sham-controlled, multicentre REVITA-2 feasibility trial. Gut. 2022 Feb;71(2):254-264. doi: 10.1136/gutjnl-2020-323608. Epub 2021 Feb 17. PMID 33597157

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects participated in a 4-week oral antidiabetic drug (OAD) run-in period before the index procedure to confirm lack of blood glucose control in conjunction with medication compliance and nutritional counseling. All subjects were managed according to current diabetes standard of care.
Groups:
- DMR Procedure (Europe); DMR Procedure (Brazil): Subjects randomized to the DMR procedure are unblinded at 24 weeks and followed for an additional 24 weeks.
  DMR Procedure: The DMR procedure consists of hydrothermal ablation of the duodenum using the Revita System
- Sham Procedure (Europe); Sham Procedure (Brazil): Subjects are unblinded at 24 Weeks. Sham subjects given option to cross over to receive DMR treatment at 24 Weeks and followed up for additional 24 weeks. Not all patients crossed over and received DMR treatment at 24 Weeks.
  Sham Procedure: The sham procedure consists of placing the Revita Catheter into the stomach for 30 minutes and then removing it from the patient.
Period: First 24 Weeks
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil)
Started | 39 | 37 | 17 | 16
Completed | 39 | 36 | 17 | 16
Not Completed | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Second 24 Weeks (Crossover for Sham)
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil)
Started | 33 | 0 | 4 | 0
Completed | 33 | 0 | 4 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Procedure (Europe); Sham Procedure (Brazil): Subjects are unblinded at 24 Weeks. Sham subjects to cross over to receive DMR treatment at 24 Weeks and followed up for additional 24 weeks.
  Sham Procedure: The sham procedure consists of placing the Revita Catheter into the stomach for 30 minutes and then removing it from the patient.
- Total: Total of all reporting groups
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil) | Total
Number analyzed (Participants) | 39 | 36 | 17 | 16 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 16 | 13 | 86
  >=65 years | 12 | 6 | 1 | 3 | 22
Age, Continuous [Median (Full Range); unit: years] | 59 [40 to 72] | 56.5 [35 to 75] | 56 [35 to 72] | 57.6 [42 to 73] | 58 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 8 | 33
  Male | 30 | 28 | 9 | 8 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 25 | 21 | 12 | 13 | 71
  Race: Black | 0 | 0 | 4 | 3 | 7
  Race: Asian | 0 | 1 | 1 | 0 | 2
  Race: Other | 1 | 2 | 0 | 0 | 3
  Race: undisclosed | 13 | 12 | 0 | 0 | 25
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 9 | 0 | 0 | 17
  Belgium | 9 | 7 | 0 | 0 | 16
  Brazil | 0 | 0 | 17 | 16 | 33
  United Kingdom | 11 | 12 | 0 | 0 | 23
  Italy | 11 | 8 | 0 | 0 | 19
BMI (kg/m2) [Median (Full Range); unit: kg/m2] | 31.4 [23.6 to 39.5] | 30.4 [24.2 to 39.6] | 32.3 [25.5 to 37.4] | 31.6 [26.1 to 37.9] | 31.4 [23.6 to 39.6]
Fasting Glucose [Median (Full Range); unit: mg/dL] | 191 [122 to 313] | 185 [110 to 344] | 190 [141 to 289] | 182 [119 to 263] | 187 [110 to 344]
HbA1c (%) [Median (Full Range); unit: % of glycosylated hemoglobin] | 8.1 [7.5 to 10] | 8.2 [7.5 to 10] | 8.6 [7.5 to 9.6] | 8.15 [7.5 to 9.4] | 8.26 [7.5 to 10]
MRI-PDFF (%) among subjects with baseline MRI-PDFF >5% [Median (Full Range); unit: % of liver fat] | 16.46 [5.47 to 32.98] | 16.11 [5.58 to 35.75] | 16.45 [6.96 to 31.76] | 16.98 [6.95 to 33.88] | 16.5 [5.47 to 35.75]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 24 Weeks in Hemoglobin A1c (HbA1c), DMR vs Sham.
Description: The primary efficacy endpoint is the change from baseline at 24 weeks in HbA1c, DMR vs Sham
Time Frame: Baseline and 24 Weeks post-procedure
Population: mITT population
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil)
Number analyzed (Participants) | 39 | 36 | 17 | 16
percentage change from baseline | -0.60 [-1.40 to 0.20] | -0.30 [-0.80 to 0.20] | -1.85 [-2.40 to -1.10] | -1.60 [-2.00 to -1.10]

2. Primary Outcome: Change From Baseline at 12 Weeks in MR-PDFF, DMR vs Sham
Description: The absolute change from baseline at 12 weeks in MR-PDFF in patients with baseline MR-PDFF > 5% , DMR vs Sham
Time Frame: Baseline and 12 Weeks post-procedure
Population: mITT population; not all patients from participant flow were able to undergo a MRI-PDFF. All patients who had a MRI-PDFF performed are analyzed and represented below.
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil)
Number analyzed (Participants) | 33 | 28 | 15 | 15
percentage change from baseline | -5.4 [-8.35 to -2.25] | -2.24 [-4.61 to -0.32] | -5.4 [-12 to -2.84] | -6.07 [-10.95 to -3.12]

ADVERSE EVENTS:
Time Frame: Adverse events for subjects randomized to DMR (and all training cases) were followed for up to a maximum of 56 weeks. Adverse events for subjects randomized to sham who crossed-over to DMR at 24 weeks were followed for up to a maximum of 56 weeks.
Groups:
- Sham Crossover (Europe): Subjects that were in sham arm (Europe) until 24 weeks and then crossover to receive DMR treatment at 24 weeks and followed up for additional 24 weeks. AEs captured from time of DMR procedure through follow up to end of study.
- Sham Crossover (Brazil): Subjects that were in sham arm (Brazil) until 24 weeks and then crossover to receive DMR treatment at 24 weeks and followed up for additional 24 weeks. AEs captured from time of DMR procedure through follow up to end of study.
Arm/Group | DMR Procedure (Europe) | Sham Procedure (Europe) | DMR Procedure (Brazil) | Sham Procedure (Brazil) | Sham Crossover (Europe) | Sham Crossover (Brazil)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37 | 0/17 | 0/16 | 0/33 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/39 | 1/37 | 3/17 | 0/16 | 0/33 | 0/4
Other Adverse Events (participants affected / at risk) | 31/39 | 26/37 | 16/17 | 14/16 | 26/33 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DMR Procedure (Europe) (N=39) | Sham Procedure (Europe) (N=37) | DMR Procedure (Brazil) (N=17) | Sham Procedure (Brazil) (N=16) | Sham Crossover (Europe) (N=33) | Sham Crossover (Brazil) (N=4)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DMR Procedure (Europe) (N=39) | Sham Procedure (Europe) (N=37) | DMR Procedure (Brazil) (N=17) | Sham Procedure (Brazil) (N=16) | Sham Crossover (Europe) (N=33) | Sham Crossover (Brazil) (N=4)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4) | 5 (5) | 0 (0) | 3 (5) | 0 (0)
Iron Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (4) | 2 (2) | 8 (9) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (8) | 2 (2) | 1 (1) | 5 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
duodenitis (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 5 (6) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (16) | 7 (13) | 11 (106) | 12 (107) | 4 (10) | 2 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (36) | 4 (11) | 0 (0) | 0 (0) | 6 (11) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Results from prespecified interaction testing and clinical parameter assessment showed heterogeneity between European (DMR N=39; sham N=37) and Brazilian (DMR N=17; sham N=16) populations, therefore, results were stratified by region. Limitations of this feasibility study include the relatively small patient population and heterogeneity between European and Brazilian populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT02879383/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT02879383/SAP_001.pdf